CLINICAL TRIAL: NCT01533519
Title: A Dose Escalation Study of Intranasal Neuropeptide Y in PTSD
Brief Title: A Dose Escalation Study of Intranasal Neuropeptide Y in Post Traumatic Stress Disorder (PTSD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: James Murrough (Other)
Responsible Party: Sponsor-Investigator, James Murrough, Assistant Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: GCO 11-1487
Record Dates: First submitted 2012-01-31; First posted 2012-02-15 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Posttraumatic Stress Disorder
Keywords: Neuropeptide Y; Intranasal Administration; PTSD; Trauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Neuropeptide Y

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NPY/placebo (Experimental): This arm gets NPY first then placebo (saline). The placebo is 0.9% USP-grade saline without NPY.
  Interventions: Drug: Neuropeptide Y
- placebo/NPY (Experimental): This arm gets placebo (saline) first then NPY.
  Interventions: Drug: Neuropeptide Y

INTERVENTIONS:
Drug: Neuropeptide Y — Intranasal administration will be administered with a nasal drug delivery device.
  Other Names: NPY

SUMMARY:
This study is designed to investigate the safety of intranasal administration of NPY using a dose escalation, randomized, double-blinded, placebo-controlled crossover design in a medication-free, symptomatic PTSD group.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, age 18-60.
* Participants must have a level of understanding sufficient to agree to all tests and examinations required by the protocol and must sign a written informed consent document. We determine whether they have a sufficient understanding of the study procedures and risks by asking them to explain what's involved in the study and to give examples of study risks and benefits.
* Participants must fulfill DSM-IV criteria for current PTSD, based on the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I) and on the Clinician-Administered PTSD Scale (CAPS).
* CAPS score must be at least 40 (moderate PTSD severity) at screening.

Exclusion Criteria:

* Current, primary Axis I disorders other than PTSD.
* History or current bipolar disorder or primary psychotic disorders (e.g. schizophrenia, schizoaffective disorder).
* Current diagnosis of anorexia nervosa or bulimia nervosa.
* Women who are pregnant or are breast-feeding.
* Drug or alcohol abuse or dependence within the preceding 3 months.
* poorly controlled hypertension (manifest by SBP > 140 and/or DBP > 90); HR < 60 or > 100 at rest at the time of screening and confirmed immediately prior to randomization
* Evidence of coronary artery disease as evidenced by history, abnormal ECG, typical symptoms
* History of arrhythmia, cardiac surgery, or family history of sudden death
* Hepatic dysfunction as defined by AST and ALT > 2x URL, or alkaline phosphatase and bilirubin > 1.5 x URL within X days prior to randomization
* Chronic renal disease as defined by serum creatinine > 1.9
* Any other serious or unstable clinically significant abnormal findings of laboratory parameters, physical examination, or ECG as determined by the PI.
* Any other serious or unstable condition that would put the subjects at undue risk as determined by the PI or additional safety monitor.
* Serious and imminent suicidal or homicidal risk.
* Psychotropic medication that will not be tapered off at least 7 days prior to screening; withdrawal symptoms must be absent at the time of screening
* History of nasal disorders or sinonasal surgery, or significant nasal abnormalities based on nasal exam.
* Received investigational intervention within 30 days prior to randomization

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-12; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Patient Rated Inventory of Side Effects (PRISE) | baseline and within 2 hours of administration of NPY
  Clinician-administered and safety measures will take place right before and after the administration to identify and evaluate the tolerability of each possible symptom (from baseline to within 2 hours of NPY administration).

SECONDARY OUTCOMES:
State-Trait Anxiety Inventory (STAI) | baseline and within 2 hours of administration of NPY
  Self-report behavioral measures will take place right before and after the administration to evaluate acute anxiolytic effects of intranasal administration of NPY
Change in Beck Anxiety Inventory (BAI) | at baseline and within 2 hours of administration of NPY
  Self-report behavioral measures will take place right before and after the administration to evaluate acute anxiolytic effects of intranasal administration of NPY

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

REFERENCES:
- [Derived] Sayed S, Van Dam NT, Horn SR, Kautz MM, Parides M, Costi S, Collins KA, Iacoviello B, Iosifescu DV, Mathe AA, Southwick SM, Feder A, Charney DS, Murrough JW. A Randomized Dose-Ranging Study of Neuropeptide Y in Patients with Posttraumatic Stress Disorder. Int J Neuropsychopharmacol. 2018 Jan 1;21(1):3-11. doi: 10.1093/ijnp/pyx109. PMID 29186416